CLINICAL TRIAL: NCT06009666
Title: Elastographic and Ultrasonographic Evaluation of Patients With Breast Cancer Related Lymphedema and Investigation of the Relationship of These Parameters With Clinical Data
Brief Title: Elastographic and Ultrasonographic Evaluation of Patients With Breast Cancer Related Lymphedema
Status: Completed | Type: Observational
Sponsor: Marmara University (Other)
Responsible Party: Sponsor
Other Study IDs: 07.01.2022.145
Record Dates: First submitted 2023-02-03; First posted 2023-08-24 (Actual); Last update posted 2023-08-24 (Actual); Status verified 2023-08

CONDITIONS: Lymphedema of Upper Arm; Stiffness of Hand, Not Elsewhere Classified; Evaluations, Diagnostic Self

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Patient Group: Both Extremities of Patients With Breast Cancer Related Lymphedema
  Interventions: Diagnostic Test: Shear Wave Elastography and B Mode Ultrasonography; Diagnostic Test: Quick Dash Questionnare; Diagnostic Test: The Lymphedema Life Impact Scale; Diagnostic Test: Questioning lymphedema-related symptoms; Other: Extremity circumference and volume measurement
- Control Group: Both Extremities of Healthy People With No History of Breast Cancer
  Interventions: Diagnostic Test: Shear Wave Elastography and B Mode Ultrasonography

INTERVENTIONS:
Diagnostic Test: Shear Wave Elastography and B Mode Ultrasonography — We evaluated the both upper extremities of the patient and control group with elastography and B mode ultrasonography. Shear wave elastography evaluates tissue deformation caused by acoustic radiation force. A highly focused ultrasound radiation is produced; The propagation speed of the shear wave depends on the stiffness of the tissue. It is a simple, inexpensive, bedside, widely available, non-invasive technique. B mode USG can be used to assess skin and subcutaneous tissue thickness and echogenicity. Skin and subcutaneous thickness were measured with b mode ultrasound. Skin and subcutaneous tissue stiffness was measured by shear wave ultrasonography
Diagnostic Test: Quick Dash Questionnare — Quick-DASH is an assessment questionnaire that measures activity and participation limitations in all upper extremity disorders. In the questionnaire, the difficulties of the patients during their daily living activities are questioned with 11 questions. Each answer is scored from 1 to 5 on a Likert scale, from best to worst.
  Groups: Patient Group
Diagnostic Test: The Lymphedema Life Impact Scale — The Lymphedema Life Impact Scale is a questionnaire developed to evaluate the physical, functional and psychosocial effects of lymphedema. It consists of 18 questions; It includes 8 physical, 4 psychosocial and 6 functional subgroups. Each question is scored from 1 to 5, with higher scores indicating increased seriousness.
  Groups: Patient Group
Diagnostic Test: Questioning lymphedema-related symptoms — Arm pain and feeling of tension, heaviness and stiffness in the arm were evaluated separately by numerical scale. This scale is a 10 cm ruler that writes no pain, no tension, no heaviness, no stiffness on one side, and unbearable pain, tension and heaviness on the other side. Patients were asked to rate their associated symptoms on this scale between 0 and 10.
  Groups: Patient Group
Other: Extremity circumference and volume measurement — For the diagnosis of lymphedema, a detailed physical examination and extremity circumference were measured. This measurement was taken from both wrists to arm height with 4 cm intervals. Those with a circumference difference greater than 2 cm and/or no 10% volume difference were considered preclinical (latent) and those with clinical lymphedema.
  Groups: Patient Group

SUMMARY:
The aim of this study is to evaluate the feasibility of shear-wave elastography for the diagnosis and staging of breast cancer related lymphedema by assessing the skin and subcutaneous tissues of the arm and forearm, which could serve as a reference standard and be more easily applicable in daily life; and to investigate the relationship between the patients' symptoms and elastographic measurements.

DETAILED DESCRIPTION:
Both upper extremities of 72 patients with lymphedema and 72 healthy upper extremities were included in the study. The patients' demographic and clinical data were recorded. The thickness and echogenicity of the skin and subcutaneous tissues of all extremities were evaluated with B-mode ultrasonography, and the stiffness of the skin and subcutaneous tissues was evaluated with shear-wave elastography. The lymphedema arm and the healthy arm of the patients were compared both with each other and with the data of the control group. Interobserver and intraobserver reliability analysis was performed for ultrasonography and elastography measurements. The patients' pain, tension, weight, and stiffness symptoms associated with lymphedema were questioned using a numerical scale. The patients' functionality and participation in daily life activities were evaluated with the Quick DASH and Life Impact Index questionnaires. The relationship between these findings and elastographic and ultrasonographic parameters was analyzed.

ELIGIBILITY:
Inclusion Criteria:

For the patient group

* between the ages of 18-75
* diagnosed with breast cancer-associated lymphedema by lymphoscintigraphy
* being stage 0-1-2 lymphedema according to ISL staging For the control group
* between the ages of 18-75
* no history of breast cancer

Exclusion Criteria:

* History of surgery in the assessment area
* History of trauma at the assessment site
* Active infection in the assessment area
* Presence of congenital or acquired malformations at the assessment site
* Primary lymphedema
* those with any medical condition that may cause edema, such as advanced heart or kidney failure

Ages: 18 Years to 75 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: In our study, individuals with breast cancer-related lymphedema diagnosis followed by Marmara University Pendik Training and Research Hospital Physical Medicine and Rehabilitation Department were included in the patient group, while upper extremity data of healthy volunteers without a known lymphedema history were controlled by one-to-one matching, considering the dominant and lymphedema sides of the patient group. included in the group.
Sampling Method: Non-Probability Sample
Enrollment: 72 (Actual)
Dates: Start 2022-02-01 (Actual); Primary Completion 2022-04-01 (Actual); Study Completion 2022-11-01 (Actual)

PRIMARY OUTCOMES:
B Mode Ultrasonography Measurements | Day 0
  Arm and forearm skin and subcutaneous tissue thicknesses in milimetres evaluated by B mode USG
Shear Wave Elastography Measurements | Day 0
  Arm and forearm skin and subcutaneous tissue stiffness in kilopascal evaluated by Shear wave elastography
B Mode Ultrasonography Measurements | Day 0
  Arm and forearm skin and subcutaneous tissue SEG and SEFS grades evaluated in echogenicity grade system by B mode USG

SECONDARY OUTCOMES:
Association of USG and SWE Measurements With Symptoms | Day 0
  It is the relationship between the parameters evaluated by USG ( thickness in milimetres echogenity according to grading system) and SWE (stiffness in kilopascal) and the pain, tension, heaviness and stiffness scoring in which symptoms in numeric scale.
Association of USG and SWE Measurements With Functionality | Day 0
  It is the relationship between the parameters evaluated by USG (thickhickness in milimetres , echogenity according to grading system) and SWE (stiffness in kilopascal) and QUİCK DASH Questionnaire Score
Association of USG and SWE Measurements With Participation İn Daily Life | Day 0
  It is the relationship between the parameters evaluated by USG (thickness in milimetres ,echogenity according to grading system) and SWE (stiffness in kilopascal) and The Life İmpact Questionnaire Scale
Association of USG and SWE Measurements With Volume Measurements | Day 0
  It is the volume measurement of both arms of the patients in cubic centimetre.

CONTACTS AND LOCATIONS:
Overall Officials: CANAN ŞANAL TOPRAK, Study Chair — Marmara University
Locations (2):
- Turkey (Türkiye) (2):
  - Canan Şanal-Toprak, Istanbul
  - Marmara University School of Medicine, Pendik Education and Research Hospital, Department of Physical Medicine and Rehabilitation, Istanbul

IPD SHARING:
Plan to Share IPD: Undecided